CLINICAL TRIAL: NCT06881693
Title: Optimizing Therapist-guided Internet-delivered Cognitive Behaviour Therapy for New and Expecting Parents
Brief Title: Internet-Delivered Cognitive Behaviour Therapy for Depression and Anxiety in Perinatal Parents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Government of Saskatchewan, Ministry of Health (Unknown); Macquarie University, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 985
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Anxiety; Depression
Keywords: Anxiety; Depression; Internet-delivered cognitive behaviour therapy; Patient stories; Perinatal mental health
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: All clients will be directed to complete the Wellbeing Course for New and Expecting Parents
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wellbeing Course for New and Expecting Parents (Experimental): Participants in the current study will be perinatal parents experiencing symptoms of depression and/or anxiety. All participants will have access to 5 ICBT lessons released gradually over 8 weeks. The 5 ICBT lessons target challenges and symptoms of anxiety and depression in perinatal parents and focus on: 1) symptom identification and the cognitive behavioural model; 2) thought monitoring and challenging; 3) de-arousal strategies and pleasant activity scheduling; 4) graduated exposure; and 5) relapse prevention. Materials are text-based with visual images, and are presented as slideshows, stories, homework reflections, and additional resources.
  Interventions: Behavioral: Internet-delivered Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Internet-delivered Cognitive Behavioural Therapy — The Wellbeing Course for New and Expecting Parents (WCNEP) is an adaptation of the Wellbeing Course (developed and evaluated at Macquaire University, Australia) and the Wellbeing Course for New Moms (a Canadian adaptation of the Wellbeing Course for new moms). The WCNEP is a transdiagnostic ICBT intervention designed for perinatal parents experiencing depression and/or anxiety, and will be offered by the Online Therapy Unit, a unit providing routine care ICBT services in Canada. The WCNEP will be evaluated in phases; phase 1 will evaluate the course for birthing parents only and phase 2 will evaluate the course for birthing and non-birthing parents. Therapist support will be offered for 8 weeks, with the possibility to extend the support to 12 weeks. Therapists will spend ~15 minutes/week communicating with each client, via secure messages. Phone calls will only be made if there is a significant clinical issue requiring attention that the therapist feel cannot be addressed in messages.

SUMMARY:
This study evaluates the effectiveness of the Wellbeing Course for New and Expecting Parents (WCNEP), an internet-delivered cognitive behavioral therapy (ICBT) intervention, in reducing symptoms of anxiety and depression in perinatal parents, within a routine care online therapy clinic (the Online Therapy Unit). The study aims to assess treatment uptake, perceptions, feasibility, and effectiveness of the WCNEP in routine care among birthing and non-birthing parents. Over the duration of 8 weeks, participants will review course materials online and respond to questionnaires aimed at assessing changes in various outcomes over time.

DETAILED DESCRIPTION:
Depression and anxiety in the perinatal stage are associated with adverse outcomes such as pregnancy and birth complications, developmental impacts on the baby, relationship issues and poor wellbeing with the partner. Despite these challenges, barriers such as stigma and shame, poor understanding and awareness of symptoms, and lack of treatment availability prevent access to treatment.

Internet-delivered cognitive behaviour therapy (ICBT) is an effective and accessible treatment. The Online Therapy Unit (OTU) routinely delivers ICBT programs for various concerns to Saskatchewan residents. ICBT programs offered by OTU have shown great success, particularly in addressing symptoms of depression and anxiety. Furthermore, previous trials conducted by OTU - Maternal Depression Online and Wellbeing Course for New Moms - have demonstrated the effectiveness of the programs in addressing postnatal depression and anxiety among birthing parents.

Despite the effectiveness of these programs, they were limited in scope; Maternal Depression Online was primarily designed to address depression, and both programs were offered exclusively to postnatal birthing parents. Accordingly, the Wellbeing Course for New and Expecting Parents (WCNEP) has been developed as an 8-week transdiagnostic ICBT program for perinatal birthing and non-birthing parents experiencing depression and/or anxiety. To develop the WCNEP, the Wellbeing Course for New Moms was adapted for parents across the perinatal stage by revising the program content and incorporating additional patient stories of perinatal birthing and non-birthing parents.

Although recruitment and service provision will include both birthing and non-birthing perinatal parents, the Course will be evaluated in two phases. In phase 1, the investigators will evaluate the Course for perinatal birthing parents. In phase 2, the investigators will evaluate the course for non-birthing parents. Prospective clients may learn about the WCNEP from advertisements to the public, healthcare providers, and community organizations. Interested clients will be directed to the study website to complete a screening protocol. Clients will subsequently book and complete a telephone screening with an OTU therapist. Following the telephone screening, eligible clients will be enrolled in the WCNEP. Participants will have access to five lessons that they will complete in consecutive order with 1 to 2 weeks between lessons. They will be asked to complete questionnaires at various time points, and provided with homework activities to complete after each lesson. Participants will also have access to therapist support for a minimum of 8 weeks, which can be extended up to 12 weeks in the event that the birth of a child or some unexpected event occurs during the duration of the Course. After completing treatment, a subset of participants will take part in a semi-structured interview for feedback on overall course content and specific course components (i.e., patient stories).

The overall goals of the study are to evaluate the effectiveness of the intervention on various outcomes in perinatal parents over time, and the uptake of and engagement with different components (e.g., patient stories) of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Become the guardian of an infant in the last 24 month by birth or adoption/fostering or are expecting the birth of an infant as a birthing parent or partner;
* Self-reported difficulty with depression and/or anxiety;
* Are aged 18 years or older; or 16 if participant meets criteria to be treated as a mature minor based on Saskatchewan legislation;
* Willingness to learn information and skills to self-manage mental health difficulties, consent to course and associated research.

Exclusion Criteria:

* Current severe medical or psychiatric condition that requires immediate treatment (e.g. current mania or psychosis, actively suicidal or unable to keep themselves safe, medical condition requiring immediate surgery or other invasive treatment);
* Living outside of Saskatchewan;
* Unable to read and understand English. (All content is provided in English and staff is English speaking; it is cost prohibitive at this time to provide the complete service in languages other than English).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | Baseline (Screening), weeks 1-8, and 20 weeks from enrollment
  Tracking the change in depression symptoms. 10 items are measured on a 4-point Likert scale ranging from 0-3. Scores are summed with total scores ranging from 0 to 30. Higher scores are associated with higher depression severity.
Generalized Anxiety Disorder 7-item (GAD-7) | Baseline (Screening), weeks 1-8, and 20 weeks from enrollment
  Tracking the change in anxiety symptoms. 7 items are measured on a 4-point Likert scale ranging from 0-3. Scores are summed into a total score ranging from 0 to 21, with higher scores indicating more severe self-reported levels of anxiety.

SECONDARY OUTCOMES:
Shortened Postpartum Bonding Questionnaire (S-PBQ) | Baseline (Screening), week 8 and 20 weeks from enrollment
  Tracking the change in postnatal birthing parents' bonding with their baby. 10 items are measured on a 5-point Likert scale, ranging from 1-5. Scores are summed into a total score ranging from 10 to 50, with higher scores indicating greater self-reported difficulties in bonding with baby. Administered to postnatal parents only.
UCLA 3-Item Loneliness Scale | Baseline (Screening), week 8 and 20 weeks from enrollment
  Measures loneliness. 3 items are measured on a 3-point Likert scale ranging from 1-3. Scores are summed into a total score ranging from 3 to 9, with higher scores indicating higher levels of perceived loneliness.
Multidimensional Scale of Perceived Social Support (MSPSS) | Baseline (Screening), Week 8, 20 weeks from enrollment
  A 12-item measure with three subscales measuring perceived social support from friends, family and significant other. Each subscale contains 4-items. Items on each subscale are measured on a 7-point Likert scale, ranging from 1-7. Subscale scores range from 4 to 28 each, with higher scores indicating greater perceived social support in each category. Global scores range from 12 to 84, with higher scores indicating greater perceived social support overall.
Treatment and Story Reflection Questionnaire | Weeks 2 to 8
  Measures clients' week-to-week experience in the Wellbeing Course for New and Expecting Parents, and feedback on patient stories. This 10-item measure has been developed by the research team, and contains three subscales. Three items measured on a 7-point Likert scale ranging from 1-7 will be summed into a total score between 3 to 21 to reflect engagement with the treatment, with higher scores indicating greater engagement. Four items (three measured on an 8-point Likert scale ranging from 0-7, and one measured on a 6-point Likert scale ranging from 0-5) will be summed into a total score between 0 to 26 to reflect engagement with patient stories over the past week. Higher scores indicate greater engagement with patient stories. The remaining three items do not have a sum scores, and are used to inquire about which lesson and resources clients worked on, and client success and challenges over the previous week.
Treatment Satisfaction Questionnaire | Week 8
  A 15-item questionnaire used to assess satisfaction with treatment and negative effects experienced by clients during treatment. The questionnaire utilizes a combination of Likert-scale (5-point (0-4)and 6-point (0-5) ), open-ended, and dichotomous yes/no response options to gauge participants' perception of the course. The questionnaire has been developed by the research team and does not have scoring at this time.
Additional Resources Questionnaire | Week 8
  A 4-item measure of clients' opinions of and satisfaction with the 11 additional resources offered alongside the Wellbeing Course for New and Expecting Parents. The questionnaire utilizes a combination of dichotomous yes/no (1-item), checklist (2-items), and open-ended (1-item) response option to understand which additional resources participants reviewed and their perception of the resources. The questionnaire was developed by the research team and no score is calculated or created.
Credibility/Expectancy Questionnaire (CEQ) | Baseline (Screening) and week 4
  Measures treatment credibility and expectancy using 6 items, with two subscales. Each subscale contains 3-items. The first three items of the scale (credibility subscale) are measured on a 1-9 point Likert scale, with scores ranging from 3 to 27 on this subscale. The three items of the expectancy subscale are measured on a 9-point Likert scale ranging from 1 to 9. These items are summed to produce a subscale score ranging from 1 to 27. Higher scores in each sub-scale indicate greater treatment credibility or treatment expectancy respectively.
Semi-Structured Interview | After week 8
  A semi-structured interview to gather feedback on the treatment and specific treatment components (i.e., patient stories). The number of participants to be interviewed will be determined based on the saturation of themes yielded within preliminary qualitative analyses. The semi-structured interview questions were developed by the research team.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- Online Therapy Unit, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to the primary unit running the study — https://www.onlinetherapyuser.ca/